CLINICAL TRIAL: NCT02341430
Title: A Longitudinal Prospective Outcomes Study of Laparoscopic Abdominal Wall Hernia Repair Using Symbotex™ Composite Mesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anne Arundel Health System Research Institute (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 689069
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Grade I Ventral Hernia; Grade II Ventral Hernia
Keywords: hernia; synthetic mesh
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Symbotex™ Composite Mesh — Repair of a Grade I or II ventral hernia according to VHWG classification system with Symbotex™ Composite Mesh

SUMMARY:
This study is being done to test the efficacy of Symbotex™ as an effective synthetic mesh option in the repair of grade I and II ventral hernias.

DETAILED DESCRIPTION:
This study is being done to validate the efficacy of Symbotex™ as an effective synthetic mesh option in the repair of grade I and II ventral hernias. It will also set the groundwork for a future clinical trial in which the efficacy of Symbotex® can be compared to other synthetic mesh products on the market.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Grade I or II ventral hernia according to VHWG classification system
* Pre-operative informed consent is obtainable

Exclusion Criteria:

* Not candidate for laparoscopic approach for repair of their hernia
* Determination in the operating room that biologic mesh is needed over permanent mesh
* Fascial defect less than 3 cm in greatest dimension
* Concurrent placement of another mesh (synthetic or biologic ) at the site where the study mesh is placed
* Grade III or IV ventral hernia according to VHWG system
* ASA score IV or above
* Any disease or condition along with the surgeon's clinical judgment that contraindicates the use of study mesh. These include but are not limited to the presence of chronically infected tissues subjecting patient to risk of synthetic mesh infection, accidental bowel injury during surgery or anatomy of the patient that is not receptive to laparoscopic surgery or mesh implantation.
* Pregnancy
* Use of more than one of the same study mesh is not an exclusion criterion in and of itself, so long as the type of mesh is selected according to the randomization protocol. In other words, if the hernia defect is larger than the largest Symbotex™ mesh available, two or more Symbotex mesh pieces may be used to appropriately repair the hernia defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Hernia Recurrence | One year
Quality of Life | One year
Hernia associated pain and movement limitations pre-surgery compared to post-surgery | One year
Reoperation Rate | One year
Percutaneous Intervention Rate | One year
Number of Participants with Adverse Events as a Measure of Safety and Tolerability" | One year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Park, M.D., Principal Investigator — Anne Arundel Medical Center
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

REFERENCES:
- [Background] Ventral Hernia Working Group; Breuing K, Butler CE, Ferzoco S, Franz M, Hultman CS, Kilbridge JF, Rosen M, Silverman RP, Vargo D. Incisional ventral hernias: review of the literature and recommendations regarding the grading and technique of repair. Surgery. 2010 Sep;148(3):544-58. doi: 10.1016/j.surg.2010.01.008. Epub 2010 Mar 20. PMID 20304452
- [Background] Heniford BT, Park A, Ramshaw BJ, Voeller G. Laparoscopic repair of ventral hernias: nine years' experience with 850 consecutive hernias. Ann Surg. 2003 Sep;238(3):391-9; discussion 399-400. doi: 10.1097/01.sla.0000086662.49499.ab. PMID 14501505
- [Background] SymbotexTM clinging effect observed during the design validation conducted by Covidien in porcine model in May 2013- covidien internal memorandum 0901CR261a (July 2013)
- [Background] Malangoni MA and Rosen MJ. Chapter 46: Hernias, Sabiston Textbook of Surgery 19th Edition. Elsevier; Philadelphia, PA. 2012: 1128-1135
- [Background] Heniford BT, Walters AL, Lincourt AE, Novitsky YW, Hope WW, Kercher KW. Comparison of generic versus specific quality-of-life scales for mesh hernia repairs. J Am Coll Surg. 2008 Apr;206(4):638-44. doi: 10.1016/j.jamcollsurg.2007.11.025. Epub 2008 Feb 1. PMID 18387468
- [Background] Itani KM, Hur K, Kim LT, Anthony T, Berger DH, Reda D, Neumayer L; Veterans Affairs Ventral Incisional Hernia Investigators. Comparison of laparoscopic and open repair with mesh for the treatment of ventral incisional hernia: a randomized trial. Arch Surg. 2010 Apr;145(4):322-8; discussion 328. doi: 10.1001/archsurg.2010.18. PMID 20404280